CLINICAL TRIAL: NCT03262636
Title: Two-Part Study to Evaluate the Safety and Efficacy of Image Guided Surgery Using Indocyanine Green for Intramolecular Imaging of Nervous System Tumors Compared to Standard of Care, (TumorGlow)
Acronym: TumorGlow(TM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0822231
Record Dates: First submitted 2016-09-06; First posted 2017-08-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor, Primary; Brain Tumor, Recurrent
MeSH Terms: conditions — Brain Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diagnostic value of Second Window ICG (Other): The primary study objective is to determine the diagnostic value of Second Window ICG (delayed, high dose IV administration of ICG) in the surgical resection of nervous system tumors.
  The first objective is to determine safety/efficacy of high dose, delayed indocyanine green (second window ICG) during surgery of nervous system tumors.
  Interventions: Drug: Indocyanine Green
- Optimal timing and dose of SWG (Other): The second study objective is to calculate diagnostic test characteristics (sensitivity/specificity) of delayed, high dose indocyanine green (second window ICG) as a diagnostic aid during surgery of nervous system tumors.
  The third study objective is to optimize timing and dose of second window Indocyanine Green during surgery of nervous system tumors, based on sensitivity/specificity.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Indocyanine Green
  Other Names: ICG

SUMMARY:
Primary malignant and non-malignant brain tumors account for an estimated 21.42 cases per 100,000 for a total count of 343,175 incident tumors based on worldwide population estimates [1]. These entities result in variable but disappointing rates of survival, particularly for primary brain tumors (5-year survival rates: anaplastic astrocytoma 27%; glioblastoma multiforme 5%) [2, 3]. Metastatic brain tumors outnumber primary brain tumors (estimates as high as 10:1) as they affect approximately 25% of patients diagnosed with cancer [4-6]. In terms of brain tumor surgery, the extent of surgical resection-a factor that is greatly impacted by a Neurosurgeon's ability to visualize these tumors-is directly associated with patient outcomes and survival [7-9]. Although spinal cord tumors are lower in terms of their incidence [10], data correlating extent-of-resection to outcomes and survival have been demonstrated in patients with intramedullary tumors [11].

Using systemically delivered compounds with a high sensitivity of detection by near-infrared (NIR) fluorescence, it would be possible for us to improve surgical resection thus minimizing chances of recurrence and improving survival. Simply, if the tumor cells will "glow" during surgery, the surgeons are more likely to identify tumor margins and residual disease, and are, therefore more likely to perform a superior cancer operation. By ensuring a negative margin through NIR imagery, it would make it possible to decrease the rates of recurrence and thus improve overall survival.

This concept of intraoperative molecular imaging requires two innovations:

(i) a fluorescent contrast agent that can be injected systemically into the subject and that selectively accumulates in the tumor tissues, and (ii) an imaging system that can detect and quantify the contrast agent in the tumor tissues.[12, 13]

Subjects undergo intraoperative imaging, receiving an injection of indocyanine green and then undergoing intraoperative imaging of the surgery site with a NIR imaging system. The imaging devices allow the operating field to be observed in real-time.

DETAILED DESCRIPTION:
Indocyanine green is a water-soluble tricarbocyanine dye routinely used in clinical settings for measuring cardiac output, hepatic function, liver blood flow and ophthalmic angiography and has been in use for over 60 years [14]. This protocol utilizes Patheon's indocyanine green, NDC 17238-424. The chemical formula is C45H47N2O6S2Na and the compound has a molecular weight of 774.96Da (CAS number 3599-32-4). It has a peak absorption in the NIR spectrum at 800nm and maximal emission at 835nm. Indocyanine green is rapidly and completely bound to plasma proteins (especially albumin) after intravenous (IV) injection in the blood [15].

Indocyanine Green for Injection USP is a sterile, lyophilized green powder containing 25 mg of indocyanine green with no more than 5% sodium iodide. It is packaged with Sterile Water for Injection, USP, which is used to dissolve the indocyanine green, and is to be administered intravenously

ELIGIBILITY:
Inclusion Criteria

1. Adult patients 18 years of age and older.
2. Patients presenting with a CNS tumor presumed to be resectable and are at risk for local recurrence on pre-operative assessment
3. Good operative candidate as determined by the treating physician and multidisciplinary team
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria

1. Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery
2. Subjects with a history of iodide allergies
3. Vulnerable patient populations

   a. Patients unable to participate in the consent process (children and neonates).
4. Patients with non-MRI compatible implanted metallic foreign bodies are excluded from this study"
5. Patients who due to severe claustrophobia cannot tolerate MRI scanning"
6. Patients with a known allergy or hypersensitivity to MRI contrast agents including gadolinium .
7. Patients with moderate to end-stage renal (kidney) disease, defined as a glomerular filtration rate (GFR) less than 30 mL/day/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2015-06; Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Determining the sensitivity of ICG uptake and expression in identifying ANS tumor deposits when excited by an imaging probe. | 36 months

SECONDARY OUTCOMES:
optimize timing and dose of second window Indocyanine Green during surgery of nervous system tumors, based on sensitivity/specificity. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: John Y.K. Lee, MD, Principal Investigator — UPENN Neurosurgery

REFERENCES:
- [Result] Ostrom QT, Gittleman H, Liao P, Rouse C, Chen Y, Dowling J, Wolinsky Y, Kruchko C, Barnholtz-Sloan J. CBTRUS statistical report: primary brain and central nervous system tumors diagnosed in the United States in 2007-2011. Neuro Oncol. 2014 Oct;16 Suppl 4(Suppl 4):iv1-63. doi: 10.1093/neuonc/nou223. No abstract available. PMID 25304271
- [Derived] Li C, Buch L, Cho S, Lee JYK. Near-infrared intraoperative molecular imaging with conventional neurosurgical microscope can be improved with narrow band "boost" excitation. Acta Neurochir (Wien). 2019 Nov;161(11):2311-2318. doi: 10.1007/s00701-019-04054-5. Epub 2019 Sep 3. PMID 31482242